CLINICAL TRIAL: NCT03027830
Title: Physiological and Clinical Assessment of the Provisional Side-branch Intervention Strategy for Coronary Bifurcation Lesions Using iFR Pressure Wires
Brief Title: iFR Pressure Wires in Assessment of the Provisional Side-branch Intervention Strategy for Bifurcation Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova-Med Medical Research Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Bifurcation Lesions
Keywords: Provisional side-branch intervention strategy; iFR; Pilot study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iFR pressure-wire (Experimental)
  Interventions: Device: iFR pressure-wire
- Conventional (Active Comparator)
  Interventions: Device: Conventional

INTERVENTIONS:
Device: iFR pressure-wire — The instantaneous wave-free ratio (iFR) as an adenosine-independent index of coronary stenosis severity, calculated as the ratio between the distal trans-stenotic pressure and the proximal coronary pressure during a specific diastolic wave-free period
  Arms: iFR pressure-wire
Device: Conventional — Other diagnostic devices (including FFR and angiography)
  Arms: Conventional

SUMMARY:
Even in the era of drug-eluting stents, bifurcation lesions remain one of the most challenging lesion subsets in coronary intervention practice. This study was performed to evaluate the functional outcomes of pressure wires (IFR)-guided jailed side-branch intervention strategy.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) measurements require minimal and constant microvascular resistance which is routinely achieved by intravenous adenosine infusion. Adenosine-induced hyperemia establishes an optimal vascular environment for FFR measurement. However, breathlessness and chest tightness are common adverse events during adenosine infusion and severe asthma occurs occasionally. The Introduction of an adenosine-independent index (instantaneous wave-free ratio [iFR]) into clinical practice offered easier and hyperemia-free method for lesion assessment.

Physiological changes and clinical evaluation of iFR warrants further research. Therefore, the investigators conducted this study to evaluate the functional aspects of iFR-guided provisional jailed side-branch intervention strategy and compare clinical endpoints to conventional non-iFR-guided operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome
* Jailed side-branch of a vessel size > 2 mm
* Vessel length > 40 mm
* Lesion length < 10 mm by visual estimation

Exclusion Criteria:

* Significant stenosis in the left main coronary artery or the main branch proximal to the stented segment
* Totally occluded bifurcation lesions
* Primary myocardial disease
* Serum creatinine level of ≥ 2.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Physiological evaluation of iFR-guided intervention | 6-month
  iFR changes after drug-eluting balloon (DEB) inflation of the jailed side branch.

SECONDARY OUTCOMES:
length of hospital stay | 6-month
Procedure time | 30-day
Fluoroscopy time | 30-day
In-hospital heart failure class | 30-day
6-month heart failure class | 6-month
Post-PCI angina | 6-month
  Comparison of the incidence of angina after performing PCI in both the iFR and conventional groups
Ejection fraction at 6 months' post operation | 6-month
The amount of dye injection for angiography | 30-day

IPD SHARING:
Plan to Share IPD: No